CLINICAL TRIAL: NCT07041502
Title: Co-creation of the Aut-CARE Intervention to Improve the Cognitive and Emotional Functioning of Young Adults on the Autism Spectrum and Facilitate Their Socio-occupational Integration
Brief Title: Aut-CARE Intervention to Improve Cognitive and Emotional Functioning in Young Adults on the Autism Spectrum
Acronym: Aut-CARE
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-AUT-2024-102
Record Dates: First submitted 2025-05-30; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder; Autism Spectrum Disorder With Absence of Functional Language
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Aut-CARE — There is no intervention

SUMMARY:
Currently, many autistic youths struggle to adapt to academic programs or the workforce, often turning to third-sector organizations such as specialized associations and foundations. This may be due to factors such as emotional dysregulation and executive dysfunction, which interfere with their psychosocial adaptation abilities, leading to anxiety and depression. These challenges have a neurobiological basis tied to the unique complexities of the autistic brain, which experiences emotional and cognitive overload and lacks attentional filters. To address this issue, the emotional and executive functioning of autistic youths at the Friends Foundation will be assessed through objective and subjective assessments.

This data collection will serve as a foundation for conceptualizing and co-creating a more realistic affective-cognitive remediation program, integrating user perspectives (conceptualization of interventions for systematic implementation). The program aims to improve the socio-occupational and emotional adaptation difficulties that often contribute to mental health challenges within this underserved population. It is important to highlight that many existing programs focus on cognitive training and social skills, neglecting strategies for adaptation and emotional regulation. This project will stand out for its inclusive design, featuring a representative sample of both sexes, overcoming the usual limitation of male-centered approaches.

DETAILED DESCRIPTION:
The mixed or hybrid sequential study design (quantitative → qualitative → quantitative) includes three parts:

A) Assessment of socio-occupational, neuropsychological, and psychological variables to establish relationships between the degree of impairment and socio-occupational integration. Quantitative study.

B) Focus groups to determine the contents of the intervention program, which will be co-created as the Aut-CARE program. Qualitative study.

C) Pilot study of the Aut-CARE program to evaluate its format, content, feasibility, and acceptability.

Individuals aged 16 to 30 years with an ASD diagnosis, levels 1 and 2. The calculated sample size is 37 subjects for sub-study A; the minimum sample size for the focus groups (sub-study B) is 14; and a maximum of 10 participants for the pilot study (sub-study C).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 16 to 30 years (male, female, and non-binary)
* Attending one or more services of the Friends Foundation (Prelaboral Friends, Laboral Friends, and EducaFriends).
* Diagnosed with ASD (according to DSM-5 criteria), levels 1 or 2, and without intellectual disability (IQ > 80).

Exclusion Criteria:

* None

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals (females and males) aged 16 to 30 years with an ASD diagnosis, levels 1 and 2
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Difficulties in emotion regulation scale (DERS) | 1 day
  The DERS is a measure of emotional dysregulation. The raw scores range from 36 to 180. Higher scores mean more difficulties.
Battery of cognitive tests | 1 day
  A set of neuropsychological tests is administered: Trail Making Test-A, Trail Making Test-B, Digit Symbol Substitution Test, Digit Span, Letter and Numbers, and Phonetic Fluency (PMR). Scores will be t-transformed (mean=50, SD=10), so high scores mean better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Institut de Recerca de lHospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided